CLINICAL TRIAL: NCT05257044
Title: Acute Effects of Cannabigerol (CBG) on Mood and Cognition
Brief Title: Acute Effects of Cannabigerol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Carrie Cuttler, Assistant Professor, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19162
Record Dates: First submitted 2021-12-06; First posted 2022-02-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Focus: To Examine Acute Effects of CBG on Anxiety, Stress, and Cognition
Keywords: Anxiety, Stress, Memory, Mood, Cognition, Side Effects
MeSH Terms: conditions — Anxiety Disorders | interventions — cannabigerol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to ingest either CBG or a placebo in the first session. Those who ingest CBG in session 1 will ingest placebo in session 2. Those who ingest placebo in session 1 will ingest CBG in session 2.
Who Masked: Participant, Outcomes Assessor
Masking Description: The vials of CBG and placebo will be color-coded and only the PI will know what the color codes mean. Participants and the research assistant will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBG (Experimental): Participants will ingest 20 mg of CBG tincture in this arm
  Interventions: Drug: Cannabigerol
- Placebo (Placebo Comparator): Participants will ingest 20 mg of placebo tincture in this arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabigerol — Participants will ingest CBG and placebo in a double-blind randomized cross-over design
  Arms: CBG
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of hemp-derived cannabigerol (CBG) on anxiety, stress, mood, and cognition. Further, the severity of various side effects of CBG (sleepiness, dry mouth, dry eyes, increased appetite) will be assessed. As such, the study is focused on better understanding some of the potentially beneficial and detrimental effects of CBG on humans.

DETAILED DESCRIPTION:
Recruitment: Prospective participants aged 21+ who have experience using cannabis-based products will be recruited from our previous survey of CBG users, from a CBG distributor in Washington (WA) state, and via social media. These prospective participants will complete a brief online survey to determine they meet eligibility requirements. Specifically, to be eligible they will need to be 21+ years of age, reside in WA state, own a smartphone, have access to a private environment where they can access a computer with a webcam connected to a high-quality and stable internet, speak fluent English, be literate, have experience using cannabis-based products without serious adverse reactions, and be free of serious psychiatric disorders, neurological and other serious medical conditions, pregnancy, or breastfeeding, or use of illicit substances in past 2 months.

Pre-Study Preparation: Eligible participants will be contacted via email and will be asked to schedule a brief 10-minute Zoom meeting to discuss the study requirements and provide informed consent. During this brief Zoom call participants will be provided with the contact information of a CBG distributor in WA state so that they can obtain a small vial of CBG tincture (20 mg) and a small vial of placebo tincture that will be color-coded by the distributor and provided to participants at no cost. The researchers will not directly provide or handle the products. Rather, participants will obtain the product on their own without compensation. Participants will also be asked to download an app called DRUID the day prior to their testing session. This app is designed to assess cognitive and motor impairment. Finally, participants will be asked to abstain from using CBG or any cannabis products for at least 24 hours prior to participation in each testing session. Questions will also be solicited and answered at this time, informed consent will be provided online and then the two testing sessions will be scheduled.

Testing Session 1: Participants will be randomly assigned to ingest either the CBG tincture (20 mg) or placebo tincture orally in the first testing session. Next, they will provide a series of baseline ratings of their mood, anxiety, and stress using 0 to 10 rating scales and the State Form of the State-Trait Anxiety Inventory. They will also provide baseline ratings of levels of intoxication and potential side effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/ racing heart) using 0 to 10 rating scales.

Once all of these baseline measures have been obtained, the research assistant (RA) will ask if she can observe the participant ingesting one of the products using a double-blind procedure (vials will be color-coded and only the PI will know which color is used to code the two products). Next, participants will complete an online survey to obtain information on demographic characteristics, cannabis and CBG use patterns, depression, anxiety, and stress. This will also provide time for the CBG to take effect. After participants complete the approximately 20-minute survey they will be asked to obtain ratings of their mood, anxiety, and stress using 0 to 10 rating scales and the State Form of the State-Trait Anxiety Inventory. The investigators will also assess potential side effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/racing heart) and drug effects using 0 to 10 rating scales. Next, participants will complete the Trier Social Stress Test and then will complete ratings of their mood, anxiety, and stress using 0 to 10 rating scales and the State Form of the State-Trait Anxiety Inventory. Next, they will complete the California Verbal Learning Test II, and the cognitive and motor tests on the DRUID app. Finally, they will complete ratings of their mood, anxiety, and stress using 0 to 10 rating scales and the State Form of the State-Trait Anxiety Inventory. The investigators will also assess potential side effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/racing heart) using 0 to 10 rating scales. This entire process (completing testing session 1) will take approximately 90-minutes total.

Testing Session 2: Approximately one-week later participants will complete the second testing session which will be identical to the first testing session with the exception of the product they will ingest. Specifically, those that ingested the CBG tincture in session 1 will ingest the placebo in session 2 and those that ingested the placebo in session 1 will ingest the CBG tincture in session 2. Also, at the end of the second testing session participants will be debriefed. Completing testing session 2 will also take approximately 90-minutes total. As such completing both sessions will require a total of 3 hours.

ELIGIBILITY:
Inclusion Criteria

* 21+ years of age
* reside in Washington state
* own a smartphone
* have access to a private environment where they can access a computer with a webcam connected to a high-quality and stable internet
* speak fluent English
* be literate
* have experience using cannabis-based products without serious adverse reactions

Exclusion Criteria

* serious psychiatric disorders (e.g., psychotic disorder, bipolar disorder)
* neurological and other serious medical conditions including head injury
* pregnancy, or breastfeeding
* use of illicit substances in past 2 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified man or woman
Enrollment: 34 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Mood | Change from baseline to approx. 20 minutes after CBG/placebo use
  Participants will provide ratings of their mood using 0-10 scales
Change in Mood | Change from baseline to approx. 40 minutes after CBG/placebo use
  Participants will provide ratings of their mood using 0-10 scales
Change in Mood | Change from baseline to approx. 60 minutes after CBG/placebo use
  Participants will provide ratings of their mood using 0-10 scales
Change in Stress | Change from baseline to approx. 20 minutes after CBG/placebo use
  Participants will provide ratings of their stress using 0-10 scales
Change in Stress | Change from baseline to approx. 40 minutes after CBG/placebo use
  Participants will provide ratings of their stress using 0-10 scales
Change in Stress | Change from baseline to approx. 60 minutes after CBG/placebo use
  Participants will provide ratings of their stress using 0-10 scales
Change in Anxiety | Change from baseline to approx. 20 minutes after CBG/placebo use
  Participants will provide ratings of their anxiety using 0-10 scales and will complete the State Form of the State-Trait Anxiety Inventory
Change in Anxiety | Change from baseline to approx. 40 minutes after CBG/placebo use
  Participants will provide ratings of their anxiety using 0-10 scales and will complete the State Form of the State-Trait Anxiety Inventory
Change in Anxiety | Change from baseline to approx. 60 minutes after CBG/placebo use
  Participants will provide ratings of their anxiety using 0-10 scales and will complete the State Form of the State-Trait Anxiety Inventory

SECONDARY OUTCOMES:
Memory | Approx. 40 minutes after ingesting CBG/Placebo
  Participants will complete the California Verbal Learning Test II (alternate forms)
Psychomotor | Change from baseline to approx. 45 minutes after ingesting CBG/Placebo
  Participants will complete the DRUID app
Change in Potential Side Effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/racing heart) | Change from baseline to approx. 20 minutes after ingesting CBG/Placebo
  Participants will provide ratings of each potential side effect using 0-10 scales
Change in Potential Side Effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/racing heart) | Change from baseline to approx. 40 minutes after ingesting CBG/Placebo
  Participants will provide ratings of each potential side effect using 0-10 scales
Change in Potential Side Effects (dry mouth, dry eyes, sleepiness, increased appetite, intoxication, heart palpitations/racing heart) | Change from baseline to approx. 60 minutes after ingesting CBG/Placebo
  Participants will provide ratings of each potential side effect using 0-10 scales

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Cuttler, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified data will be retained indefinitely
Access Criteria: Researchers wanting to conduct secondary data analysis following my own publication